CLINICAL TRIAL: NCT02281656
Title: Prospective Evaluation of Reverse End to Side Anterior Interosseous Nerve to Ulnar Nerve Transfer for Severe Compressive Ulnar Neuropathy at the Elbow
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Dr Christopher Doherty (Unknown); Dr Thomas Miller (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7126
Record Dates: First submitted 2014-09-22; First posted 2014-11-03 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Severe Compressive Ulnar Nerve Neuropathy (McGowan Grade III)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse End-to-side (Experimental): Surgery: a "reverse" end-to-side AIN to ulnar nerve transfer whereby the motor branch of the ulnar is left intact and the end of the AIN nerve is coapted to the side of the ulnar motor fascicle(5,6). The advantage of this technique is it preserves the continuity of the ulnar motor branch for axons if they do eventually reinnervate the intrinsic muscles while augmenting or "babysitting" these muscles during the time period until this occurs.
  Interventions: Procedure: Surgery:ulnar nerve subcutaneous transposition without AIN to ulnar nerve transfer.
- Surgery:standard care (Active Comparator): Surgery: the anterior interosseous (AIN) to motor branch of the ulnar nerve transfer has been established as an effective means to reinnervate ulnar innervated intrinsic hand muscles (without loss of function from using the AIN) when nerve injury is too proximal for recovering axons to reach the hand by 18 months. . The procedure (surgery) is presently the standard of care
  Interventions: Procedure: Surgery:ulnar nerve transposition with AIN to ulnar nerve transfer

INTERVENTIONS:
Procedure: Surgery:ulnar nerve transposition with AIN to ulnar nerve transfer
  Other Names: experimental
  Arms: Surgery:standard care
Procedure: Surgery:ulnar nerve subcutaneous transposition without AIN to ulnar nerve transfer.
  Other Names: standard care
  Arms: Reverse End-to-side

SUMMARY:
Ulnar nerve compression at the elbow is a common problem and can significantly affect hand function in severe cases. The current, standard treatment is Ulnar nerve decompression with or without transposition (moving the ulnar nerve to a site where there is less compression). In severe compression, the clinical results after this surgery are typically poor. Distal transfers of functioning nerves (at the level of the wrist) to the compressed ulnar nerve (anterior interosseous nerve to ulnar motor fascicles) have been suggested to "supercharge" or augment hand muscles while nerve axons regenerate from the level of the elbow after decompression/transposition. In fact, this treatment is becoming widely adopted without clear evidence that it changes outcomes. The investigators propose to prospectively compare the effectiveness of ulnar nerve decompression/transposition versus decompression/transposition and distal nerve transfer.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively compare the outcomes of patients with severe (intrinsic hand muscle dysfunction) compressive ulnar neuropathy at the elbow treated with ulnar nerve decompression and subcutaneous transposition alone versus ulnar nerve decompression with subcutaneous transposition and AIN to ulnar nerve reverse end-to-side transfer. The study objectives of this project are the following: 1. To prospectively compare the clinical outcomes of patients with severe ulnar neuropathy at the elbow who receive ulnar nerve decompression with subcutaneous transposition and AIN to ulnar motor reverse end-to-side nerve transfer versus decompression and subcutaneous transposition alone. 2. To prospectively compare the electrophysiologic outcomes (nerve conduction studies and EMG) of patients with severe ulnar neuropathy at the elbow who receive ulnar nerve decompression with subcutaneous transposition and AIN to ulnar motor reverse end-to-side nerve transfer versus decompression and subcutaneous transposition alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years) with severe compressive ulnar nerve neuropathy (McGowan grade III) at the elbow who consent to either ulnar nerve decompression with transposition alone or ulnar nerve decompression with transposition plus nerve transfer.

Exclusion Criteria:

* Patients under the age of 18 and over 70.
* Patients with ulnar neuropathy at multiple anatomic locations along the course of the nerve.
* Patients with mild to moderate ulnar neuropathy (McGowan grade I and II).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
pain scores on the numeric pain rating scale | one year
  The patient-rated ulnar nerve evaluation (PRUNE)

SECONDARY OUTCOMES:
evaluation of reinnvervation of hand intrinsic muscles | one year
  Electromyography (EMG)
functional performance assessment on the numeric scale | one year
  The patient-rated ulnar nerve evaluation (PRUNE); Michigan hand outcome questionnaire

REFERENCES:
- [Background] 1. McGowan AJ. The Results of Transposition of the Ulnar Nerve for Traumatic Ulnar Neuritis. The Journal of Bone and Joint Surgery, 32B (3): 293-301, 1950. 2. Macadam SA, Gandhi R, Bezuhly M et al. Simple Decompression Versus Anterior Subcutaneous and Submuscular Transposition of the Ulnar Nerve for Cubital Tunnel Syndrome: A Meta-Analysis. Journal of Hand Surgery (Am), 33A: 1314-1324, 2008. 3. Chung KC. Treatment of Ulnar Nerve Compression at the Elbow. Journal of Hand Surgery (Am), 33A: 1625-1627, 2008. 4. Haase SC and Chung KC. Anterior Interosseous Nerve Transfer to the Motor Branch of the Ulnar Nerve for High Ulnar Nerve Injuries. Annals of Plastic Surgery, 49: 285-290, 2002. 5. Barbour J, Yee A, Kahn LC and Mackinnon SE. Supercharged End-to-Side Anterior Interosseous to Ulnar Motor Nerve Transfer for Intrinsic Musculature Reinnervation. Journal of Hand Surgery (Am), 37A: 2150-2159, 2012. 6. Kale SS, Glaus SW, Yee A et al. Reverse End-to-Side Nerve Transfer: From Animal Model to Clinical Use. Journal of Hand Surgery (Am), 36A: 1631-1639, 2011. 7. Isaacs J. Supercharged End-to-Side Nerve Transfer: Too Soon for "Prime Time"? Journal of Hand Surgery (Am), 38A: 617-618, 2013.